CLINICAL TRIAL: NCT07119541
Title: A Pilot Randomized Controlled Trial Evaluating an Alliance-Focused Dialectical Behaviour Therapy Training Intervention for Borderline Personality Disorder
Brief Title: Testing an Alliance-Focused Dialectical Behaviour Therapy Training for Borderline Personality Disorder
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: York University (Other)
Responsible Party: Principal Investigator, Tali Boritz, Assistant Professor, York University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: e2024-091
Record Dates: First submitted 2025-07-29; First posted 2025-08-13 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Borderline Personality Disorder; Emotion Dysregulation
Keywords: Dialectical Behavior Therapy; Therapeutic Alliance; Alliance Rupture and Repair; Alliance-Focused Training; Deliberate Practice
MeSH Terms: conditions — Borderline Personality Disorder

STUDY DESIGN:
Intervention Model Description: Experimental: Alliance focused DBT training plus deliberate practice Active Control: Alliance focused DBT training plus reflective practice
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alliance-Focused DBT Training plus Deliberate Practice (Experimental): Immediately receives 4 sessions of a psychotherapy training intervention to improve ability to recognize and respond to alliance ruptures in treatments with clients with borderline personality disorder.
  Interventions: Behavioral: Alliance-Focused Dialectical Behavior Therapy plus Deliberate Practice
- Alliance-Focused Training plus Reflective Practice (Training as Usual) (Active Comparator): Immediately receives 4 sessions of a psychotherapy training intervention to improve ability to recognize and respond to alliance ruptures in treatments with clients with borderline personality disorder.
  Interventions: Behavioral: Alliance-Focused Dialectical Behavior Therapy plus Reflective Practice

INTERVENTIONS:
Behavioral: Alliance-Focused Dialectical Behavior Therapy plus Deliberate Practice — The alliance-focused DBT training plus deliberate practice is a 4-session weekly intervention delivered to therapists working with individuals with borderline personality disorder or emotion dysregulation. This training intervention involves a didactic component, video analysis, and case-based learning. Deliberate practice methods (e.g., setting individualized training goals, skills coaching, feedback, and opportunities for repeated practice) will be integrated both within and between training sessions.
  Arms: Alliance-Focused DBT Training plus Deliberate Practice
Behavioral: Alliance-Focused Dialectical Behavior Therapy plus Reflective Practice — The alliance-focused DBT training plus reflective practice is a 4-session weekly intervention delivered to therapists working with individuals with borderline personality disorder or emotion dysregulation. Trainings will involve a didactic component, video analysis, and case-based learning. Reflective practice methods (i.e., thinking about past experiences to gain insight for future actions) will be integrated both within and between training sessions.
  Arms: Alliance-Focused Training plus Reflective Practice (Training as Usual)

SUMMARY:
The study evaluates the feasibility, acceptability, and effect sizes of two alliance-focused dialectical behavior therapy (DBT) training interventions to improve therapists' abilities to recognize and respond to alliance ruptures with clients with borderline personality disorder (BPD). Participants will be randomly assigned to receive either a 4-week training as usual (TAU), which include didactic training plus reflective practice (i.e., thinking about past actions to gain insight for future actions) or a 4-week didactic training plus deliberate practice training (i.e., setting individualized training goals, skills coaching, and opportunities for repeated practice with expert feedback). A pre-post design will be used to assess effect sizes for change in participants' abilities to recognize and respond to alliance ruptures. Therapist characteristics will be assessed to determine moderating effects on training outcome. Feasibility and acceptability of the training intervention will be assessed following the trainings.

DETAILED DESCRIPTION:
Borderline personality disorder is a severe psychological disorder characterized by a pattern of emotional dysregulation, interpersonal difficulties, and impulsivity. The therapeutic alliance is the cornerstone of effective psychotherapy with clients with BPD and is positively associated with treatment retention and clinical improvement. However, the therapeutic alliance in BPD treatments can be difficult to form and maintain. BPD symptoms such as emotional instability, heightened emotional reactivity, greater susceptibility to negative emotions, and interpersonal sensitivity can impact the establishment of a strong therapeutic alliance. Additionally, when clients are emotionally dysregulated or presenting with high-risk behaviors, therapists are especially vulnerable to becoming reactive and engaging in therapy-interfering behaviors that can elicit or exacerbate alliance ruptures (i.e., tension, strain, or breakdown in the therapeutic alliance). Research suggests that therapists' abilities to effectively repair alliance ruptures when they occur is critical for positive clinical outcomes in BPD treatments.

Despite the importance of alliance rupture responsiveness in BPD treatments, many of the current methods employed in psychotherapy training do not adequately develop these therapeutic skills. Psychotherapy training typically focuses on the therapeutic relationship in an unstructured, non-systematic way, using instructional or supervision-based methods despite evidence that suggests this type of passive learning is ineffective for skill development. Recent advancements in psychotherapy training have begun to focus on improving therapists' skills in navigating alliance rupture and repair, however these trainings are often time intensive and do not sufficiently target the unique client needs and therapist challenges that emerge in BPD treatments.

The primary aim of this pilot randomized controlled trial is to evaluate the feasibility, acceptability, and effect sizes of two alliance-focused DBT training interventions to improve therapists' abilities to recognize and respond to alliance ruptures with BPD clients. Additionally, we will examine whether specific therapist characteristics moderate the impact of training. Up to eighty psychotherapists will be randomly assigned to receive either a 4-week training as usual, which includes alliance-focused training plus reflective practice or a 4-week alliance-focused training plus deliberate practice training. Both trainings include the same content but employ different training methods (i.e., deliberate practice versus reflective practice). Change in skill acquisition related to recognizing and responding to alliance ruptures will be assessed based on a set of performance tasks (interpersonal facilitative skills, process recognition, emotion recognition). Therapist characteristics of emotion regulation, empathy, emotional reactivity, and humility will be assessed by self-report to determine change in emotion regulation, humility, interpersonal reactivity, and empathy, and the moderating effects of these characteristics on training outcome. Finally, participants will be asked about the feasibility and acceptability of the training interventions.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be over the age of 18
2. Participants must be regulated health professionals in Canada who are authorized to deliver psychotherapy as part of their scope of practice, or a students in training under the supervision of a regulated health professional in Canada authorized to deliver psychotherapy as part of their scope of practice.
3. Participants must currently be providing psychotherapy
4. Participants must have access to reliable internet service
5. Participants must indicate that they are available to attend the training intervention times provided
6. Participants must agree to participate in the 4 weekly training intervention
7. Participants must state willingness to comply with study procedures (i.e., to complete pre- and post-intervention research evaluations, and between training homework exercises.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2025-11-28 (Actual); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Facilitative Interpersonal Skills Task (FIS) | Administered at baseline (pre-intervention) and at 4 weeks (post-intervention).
  An 8-item video vignette task used to assess ability to respond effectively to challenging client interactions in therapy. Scores range from 56 to 280, with higher scores reflecting higher levels of facilitative interpersonal skills.

SECONDARY OUTCOMES:
Process Recognition Task (PRT) | Administered at baseline (pre-intervention) and at 4 weeks (post-intervention).
  A 12-item video vignette task used to assess ability to accurately detect alliance ruptures. Scores range from 0-12, with higher scores reflecting greater accuracy of rupture detection.
Jerusalem Facial Expressions of Emotion Task (JeFEE) - Short Version | Administered at baseline (pre-intervention) and at 4 weeks (post-intervention).
  A 28-item video vignette task used to assess ability to accurately identify emotional expression. Scores range from 0 to 28, with higher scores reflecting greater accuracy of emotion recognition.
Comprehensive Intellectual Humility Scale (CIHS) | Administered at baseline (pre-intervention) and at 4 weeks (post-intervention).
  A 22-item self-report measure used to assess intellectual humility. Scores range from 22-110, with higher score indicating greater intellectual humility.
Interpersonal Reactivity Index (IRI) | Administered at baseline (pre-intervention) and at 4 weeks (post-intervention).
  A 28-item self-report measure that assesses empathy. Scores range from 28 to 140, with higher scores reflecting greater empathy.
Emotional Reactivity Scale (ERS) | Administered at baseline (pre-intervention) and at 4 weeks (post-intervention).
  A 21-item self-report measure that assesses emotional sensitivity, intensity, and persistence. Scores range from 0 to 84, with higher scores reflecting greater emotional reactivity
Difficulties in Emotion Regulation Scale (DERS) | Administered at baseline (pre-intervention) and at 4 weeks (post-intervention).
  A 36-item self-report measure that assesses difficulties with emotion regulation. Scores range from 36 to 180, with higher scores reflecting greater difficulties in regulating emotions.
Acceptability, Feasibility, and Appropriateness Scale (AFAS) | Administered at 4 weeks (post-intervention).
  A 14-item self-report measure that assesses implementation outcomes of acceptability, feasibility, and appropriateness. Scores range from 14 to 70, with higher scores reflecting greater acceptability, feasibility, and appropriateness of the training intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Tali Boritz, Ph.D., Principal Investigator — York University
Locations (1):
- York University, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No